CLINICAL TRIAL: NCT00902447
Title: Human Blood Cell Disorders Tissue Bank
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 08-202
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Human Blood Cell Disorders; Lymphoid, Myeloid and Erythroid Proliferative Disease
Keywords: Human Blood Cell Disorders; lymphoid, myeloid and erythroid proliferative disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — cells, tissue, serum, saliva, etc
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Human Blood Cell Disorders: Human Blood Cell Disorders Tissue Bank

SUMMARY:
The Human Blood Cell Disorder Tissue Bank will provide a convenient, comprehensive source of tissue containing populations of human blood cells from patients with various types of lymphoid, myeloid, and erythroid proliferative diseases as well as other associated conditions. The tissue bank will continue to be an invaluable asset for understanding of the biology of multiple blood cell disorders involving several cell types as well as the physiology of normal cellular counterparts affected in these disorders. Internal and external investigators will be able to utilize this tissue to test hypotheses relating to the immunologic, virologic, genetic, and molecular properties of these abnormal cells as well as normal cells from normal unaffected family members or normal aged matched subjects to provide better comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Participants or participant's Legally Authorized Representatives (LAR) must be able to understand and render voluntary, written informed consent.
* Patients must be able to contribute the required amount of blood and/or tissue without compromising their well-being or care.
* Participants must be willing to be contacted again for consideration of additional studies in the future, such as a blood draw or another action (e.g., bone marrow aspiration and/or biopsy) that would be done as part of their standard of care.

Exclusion Criteria:

* Patients who are known to be anemic, with hemoglobin <8.0g/dl.
* Patients who are known to be infected with HIV.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2009-04; Primary Completion 2030-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Accumulate tissue from patients with various blood disorders, including but not restricted to lymphoproliferative, myeloproliferative, and erythroproliferative conditions. | Indefinite

SECONDARY OUTCOMES:
Develop a database of at least 10,000 subjects who have donated samples for research as well as DNA banking, and who are willing to be contacted again for consideration of additional studies in the future. | Indefinite

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Chiorazzi, M.D., Principal Investigator — Northwell Health
Locations (1):
- The Feinstein Institute for Medical Research, Manhasset, New York, United States